CLINICAL TRIAL: NCT04877665
Title: Establishing Reference Intervals for Thyroid Stimulating Hormone in Children Under the Age of Two Years
Brief Title: Establishing RIs for TSH in Children Under the Age of Two Years
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Siraj Muneer, Resident, Aga Khan University Hospital, Pakistan
Other Study IDs: 5255-Pat-ERC-18
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Hypothyroidism
Keywords: Thyroid Stimulating Hormone; Reference Interval; Children; Pakistan
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reference intervals (RIs) of thyroid-stimulating hormone (TSH) and free thyroxine (FT4) are age, assay and population specific. Currently, the age and assay-specific RIs for TSH are not available for children under two years of age. This study aimed to establish reference intervals for serum concentrations of TSH and FT4 in healthy children aged 1-24 months as per CLSI C28-A3 guidelines.

DETAILED DESCRIPTION:
A prospective cross-sectional study was conducted at the Section of Chemical Pathology, Department of Pathology and Laboratory Medicine, AKUH Karachi Pakistan, from August 2018 to March 2019 after approval from The Aga Khan University Ethics Review Committee.

Healthy children from 1 to 24 months visiting the clinical lab for serum vitamin D testing were invited to participate in the study.

Their health status was determined by asking questions related to their medical medical history after informed consent from their parents/guardian. Children with recent abnormal total leucocyte or neutrophil count in the medical record or positive microbial cultures, history of any diagnosed disease or infection, history of hospitalization during the previous four weeks, congenital hypothyroidism or transient congenital hypothyroidism, history of maternal thyroid illness, or any medications with potential influences on the thyroid function, such as amiodarone, anti-epileptic drugs, glucocorticoids were excluded.

The RIs were established using the CLSI, C28-A3 guidelines, using a sample size of at least 120 specimens.

Serum TSH and FT4 were measured on ADVIA Centaur (Siemens Diagnostics, US), using chemiluminescence immunoassay.

The EP evaluator version 10 and SPSS version 21 were used for data analysis. Kolmogorov-Smirnov test assessed the normality of the data.

The RIs based on central 95% of the population were established. The median age of subjects, TSH and FT4 levels were calculated. For assessing differences in the male and female gender, Students' t' test was applied, taking p-value <0.050 as significant. Spearman's test computed the correlation between age, TSH and FT4 levels.

A total of 132 children were included in the study; one subject with confirmed congenital hypothyroidism (CH) was excluded from the study, shown in figure 1. The TSH and FT4 values of 131 subjects were included to establish the RIs. The median (IQR) age of the study subjects was 12 (11) months, and 78 (59.5%) were male.

Reference interval based on central 95% of the population for TSH is 0.73-4.94 µIU/mL and for FT4 is 0.81-1.51 ng/dL.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children from 1 to 24 months

Exclusion Criteria:

* recent illness, hospitalization, medication and maternal history of thyroid-related diseases, recent abnormal total leucocyte or neutrophil count in the medical record or positive microbial cultures, history of any diagnosed disease or infection, history of hospitalization during the previous four weeks, congenital hypothyroidism or transient congenital hypothyroidism, history of maternal thyroid illness, or any medications with potential influences on the thyroid function, such as amiodarone, anti-epileptic drugs, glucocorticoids

Ages: 1 Month to 24 Months | Sex: All
Age Groups: Child
Study Population: Healthy children from 1 to 24 months
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Establishing Reference Intervals for Thyroid Stimulating Hormone in Children under the age of two years | August 2018 to March 2019
  This study aimed to establish reference intervals for serum concentrations of TSH and FT4 in healthy children aged 1-24 months as per CLSI C28-A3 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Siraj Muneer, Principal Investigator — Aga Khan University
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan